CLINICAL TRIAL: NCT06104163
Title: Impact of Cantilever Design in the Posterior Areas of the Mandible on Clinical, Radiographic, and Volumetric Parameters: a Retrospective Study With 8-year Follow-up
Brief Title: Impact of Cantilever Design on Clinical, Radiographic, and Volumetric Parameters: a Retrospective Study
Status: Completed | Type: Observational
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Gaetano Isola, Researcher, University of Catania
Other Study IDs: 121-28
Record Dates: First submitted 2023-07-25; First posted 2023-10-27 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Partial Edentulism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The present retrospective study aims to evaluate the impact of cantilever design in the posterior areas of the mandible on clinical, radiographic, and volumetric parameters with an 8-year follow-up.

DETAILED DESCRIPTION:
Implant rehabilitation of posterior edentulous areas of the mandible is very complex because the presence of noble structures, such as the inferior alveolar nerve (NAI), often requires major reconstructive procedures to achieve adequate bone volume before implant placement.

To overcome these potential problems and provide patients with sufficient function and esthetics, the use of single-unit crowns (SCs) supported by implants with cantilever extensions was introduced. The length and design of cantilever extensions are associated with possible detrimental effects on implant and prosthetic survival. In light of the above, the objective of the present study is to evaluate the impact of cantilever design in the posterior areas of the mandible on clinical, radiographic, and volumetric parameters with an 8-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years;
* Patients with partial edentulism;
* Patients with systemic health or controlled medical conditions;
* Patients with healthy or treated periodontal conditions;
* Patients enrolled in regular supportive periodontal therapy (SPT);
* Patients without clinical signs of oral parafunctions (bruxism or clenching);
* Presence of 1 osteointegrated dental implant in posterior region (premolar or molar) of mandible, after transmucosal placement and healing at 3-6 months;
* Tissue level solid-screw implants with a sand-blasted and acid etched (SLA) surface with an endosseous diameter of 4.1 mm, a length of 8, 10 or 12 mm, a shoulder diameter of 4.8 mm and a supracrestal machined neck with a height of 1.8 mm (Straumann Dental Implant System, Institute Straumann AG); Use of prefabricated titanium abutments;
* Monolithic zirconia SCs manufactured by digital flow; Screwed SCs with a mesial or distal cantilever extension;
* Alternative crown design (ACD) with eccentric implant insertion, with crown-like-premolar and with distal or mesial cantilever with ovoid conformation. In the latter case, the lower abutment cross-section in the region between the crown-bridge connector mimics the shape of a root, creating an "interradicular" access route to facilitate oral hygiene maneuvers;
* Absence of occlusal contacts or guidance on the cantilever extension at baseline;
* Opposing dentition consisting of natural teeth or fixed or removable restorations;
* Availability of periapical radiography at baseline (i.e., loading of SCs) and at the analyzed timings (after 1, 3, 5, and 8 years);
* Availability of clinical measurements, such as pocket probing depth (PPD), plaque index (PI), bleeding index at probing (BOP), suppuration at probing (SUP), keratinized mucosa (KM), and mucosal recession (MR) taken at baseline (i.e., at loading of the SCs) and at 8 years after SCs loading, at four sites/implant with a Michigan graded periodontal probe (Deppeler SA); Availability of intraoral scans at baseline (i.e., at loading of the SCs) and at the analyzed time points (after 1, 3, 5, and 8 years after SCs loading) and executed using 3 Shape TRIOS 3, Germany GmbH.

Exclusion Criteria:

* Untreated or active periodontal diseases;
* Type I implant placement;
* SCs with cantilever extension replacing mandibular and maxillary incisors and canines; - - SCs with cantilever extension replacing posterior maxillary;
* SCs with cantilever extension supported by implants with a diameter ≤3.5 mm;
* SCs supported by hollow-screw and hollow-cylinder implants;
* Technical complications, such as fractures of implants, abutments, and the prosthetic artifact;
* Smoking habit (more than 15 cigarettes/day);
* Drug or alcohol abuse;
* Uncontrolled systemic diseases that could affect bone remodeling during implant osseointegration; or soft tissue healing (e.g., uncontrolled diabetes mellitus with HbA1c>7, osteoporosis);
* Use of medications that could affect bone remodeling during implant osseointegration or soft tissue healing (e.g., steroids, antiresorptive medication, radiotherapy);
* Autoimmune and/or inflammatory diseases affecting the oral cavity;
* Neurological or psychiatric handicap that could interfere with oral hygiene;
* Pregnancy or lactation periods.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with partial edentulism, treated comprehensively and continuously between 2015 and 2023, were enrolled at the School of Dentistry of the Department of General Surgery and Medical-Surgical Specialties, University of Catania, Catania, Italy, and a private outpatient regimen.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Probing Depth of the Peri-implant Pocket (PPD) | 8 years
  It is measured from the mucosal margin to the bottom of the probable peri-implant sulcus and expressed in mm.
Plaque Index (PI) | 8 years
  Evaluation of Plaque index (PI), expressed as the percentage of positive sites and measured at 4 implant sites (mesio-buccal, mesio-oral, disto-buccal and disto-oral) throught Michigan-grade periodontal probe.
Keratinized mucosa (KM) | 8 years
  Evaluation of Keratinized mucosa width (KM), measured from the restoration margin to the mucogingival junction and expressed in mm.
Mucosal recession (MR) | 8 years
  Mucosal recession (MR), of the peri-implant soft tissue, measured from the restoration margin to the mucosal margin and expressed in mm. Coronal from restoration margin is defined as (+) and apical from restoration margin defined as (-);
Bleeding and/or suppuration on probing (BOP/SUP) | 8 years
  Evaluation of Bleeding and/or suppuration on probing (BOP/SUP), within 30 seconds after probing and expressed as the percentage of positive sites and measured at 4 implantation sites (mesio-buccal, mesio-oral, disto-buccal and disto-oral).

SECONDARY OUTCOMES:
Volumetric analysis at baseline and after 8 years of follow-up | 8 years
  It was obtained by superimposing the intraoral scans of each patient, performed at baseline and eight years later through an optical scanner (3 Shape TRIOS 3 Germany GmbH), using 3D imaging software. The volumetric differences affecting the peri-implant soft tissues following prosthetic loading were expressed as a percentage and in mm3.
Radiographic examination at baseline and after 8 years of follow-up | 8 years
  All patients enrolled in the study underwent periapical radiography performed with the long parallel cone technique at baseline and 8 years after. The measure linear peri-implant marginal bone levels (BML) of single unit crowns (SCs) is the perpendicular distance, expressed in mm, from the mesial and distal edge of the implant shoulder to the first bone-to-implant contact (BIC).

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Isola, Principal Investigator — University of Catania
Locations (1):
- AOU Policlinico G. Rodolico, Catania, Italy

IPD SHARING:
Plan to Share IPD: No